CLINICAL TRIAL: NCT03086902
Title: Cryo Ablation vs. Radiofrequency Catheter Ablation for Ventricular Premature Contractions
Brief Title: Comparision of PVC Ablation Techniques
Acronym: PVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dr. Eyal Nof, Director of Invasive Electrophysiology Service, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC-3991-17
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Premature Ventricular Contraction
Keywords: Ablation; Cryo Energy; Radofrequency Ablation
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Group sample sizes of 44 in Group 1 and 44 in Group 2 achieve 80% power to detect a difference between the group proportions of -0.2000. The proportion in Group 1 (the treatment group) is assumed to be 0.2500 under the null hypothesis and 0.0500 under the alternative hypothesis. The proportion in Group 2 (the control group) is 0.2500. The test statistic used is the two-sided Z test with pooled variance. The significance level of the test was targeted at 0.0500. The significance level actually achieved by this design is 0.0531.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cryo Ablation (Experimental): PVCs will be mapped and ablated with a Cryo Ablation catheter
  Interventions: Device: Cryo Ablation catheter
- Radiofrequency Ablation (Active Comparator): In this arm PVCs will be mapped and ablated with a Radiofrequency Ablation catheter
  Interventions: Device: Radiofrequency Ablation Catheter

INTERVENTIONS:
Device: Radiofrequency Ablation Catheter — Ablation of PVC with RF energy
  Arms: Radiofrequency Ablation
Device: Cryo Ablation catheter — Ablation pf PVC with Cryo enerygy
  Arms: Cryo Ablation

SUMMARY:
Several reports have shown the utility of PVC ablation with cryo catheters. The aim of this study is to compare the outcomes and safety of Cryo vs. RF for PVCs.

DETAILED DESCRIPTION:
Background: Radiofrequency (RF) catheter ablation (CA) is an effective therapeutic strategy in eliminating refractory idiopathic ventricular outflow tract (OT) ventricular arrhythmias (VA). However, early and late recurrences occur commonly. RFCA has also been reported to be associated with collateral damage and pain. The use of Cryo ablation as a safer alternative energy source been previously described. In several reports Cryo was reported to successfully treat VA originating from the OT in the absence of ablation related pain and collateral damage to adjacent structures such as the coronaries. When comparing outcomes and complications of catheter ablation of VA from the papillary muscles of the left ventricle with either Cryo or RF, Cryo was found to be associated with significantly higher success rates and lower recurrence rates than RFCA.

Aim: To compare the outcomes and safety of Cryo vs. RF for PVCs. Methods: Patients with PVC VA will be randomized in a 1:1 fashion to RFCA or Cryo ablation. All procedures will be done using a 3-dimensional mapping system (EnSite™ NavX™ system, St. Jude Medical). Ablation will be performed at sites with earliest activation or at least pacemap exhibiting QRS morphology match of >11/12. Endpoint of procedure will be elimination and non inducibility of the clinical VA. All patients will undergo continuous monitoring for at least 12 hours post procedure and 12 lead Holter and exercise testing 1 month post procedure. Successful ablation will be defined as absence of clinical VA or > 50% reduction in arrhythmia burden on Holter in the absence of anti-arrhythmic medications.

ELIGIBILITY:
Inclusion criteria:

1. Patients referred for PVC ablation.
2. Age ≥ 18 years on a date of consent.

Exclusion criteria:

1. Contraindications for ablation
2. Serious known concomitant disease with a life expectancy of < 1 year
3. Elderly patients >80 years of age
4. Pregnancy or nursing
5. Unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of successful catheter ablation between both methods. | During procedure and 1 month follow up
  Successful ablation will be defined as absence of clinical VA or > 50% reduction in arrhythmia burden on Holter in the absence of anti-arrhythmic medication.

SECONDARY OUTCOMES:
Comparison of complications such as pericardial effusion/ tamponade, coronary artery damage and post procedure pericardial pain requiring medical management. | During Procedure
  Any complication will be assessed clinically during procedure and managed as indicated.
Comparison of procedure and fluoroscopy time between both strategies | During Procedure
  Time of procedure and fluoroscopy will be logged into CRF

IPD SHARING:
Plan to Share IPD: Undecided
All data will be kept at SMC and will be available

REFERENCES:
- [Result] Kurzidim K, Schneider HJ, Kuniss M, Sperzel J, Greiss H, Berkowitsch A, Pitschner HF. Cryocatheter ablation of right ventricular outflow tract tachycardia. J Cardiovasc Electrophysiol. 2005 Apr;16(4):366-9. doi: 10.1046/j.1540-8167.2005.40571.x. PMID 15828876
- [Result] Santangeli P, Proietti R, Di Biase L, Bai R, Natale A. Cryoablation versus radiofrequency ablation of atrioventricular nodal reentrant tachycardia. J Interv Card Electrophysiol. 2014 Mar;39(2):111-9. doi: 10.1007/s10840-013-9842-2. Epub 2013 Nov 29. PMID 24293174
- [Result] McDonnell K, Rhee E, Srivathsan K, Su W. Novel utility of cryoablation for ventricular arrhythmias arising from the left aortic cusp near the left main coronary artery: a case series. Heart Rhythm. 2014 Jan;11(1):34-8. doi: 10.1016/j.hrthm.2013.10.008. Epub 2013 Oct 3. PMID 24096170
- [Result] Chung FP, Chong E, Lin YJ, Chang SL, Lo LW, Hu YF, Tuan TC, Chao TF, Liao JN, Huang YC, Chi PC, Chan CS, Chen YY, Huang HK, Chen SA. Different characteristics and electrophysiological properties between early and late recurrences after acute successful catheter ablation of idiopathic right ventricular outflow tract arrhythmias during long-term follow-up. Heart Rhythm. 2014 Oct;11(10):1760-9. doi: 10.1016/j.hrthm.2014.06.011. Epub 2014 Jun 12. PMID 24931638
- [Result] Rivera S, Ricapito Mde L, Tomas L, Parodi J, Bardera Molina G, Banega R, Bueti P, Orosco A, Reinoso M, Caro M, Belardi D, Albina G, Giniger A, Scazzuso F. Results of Cryoenergy and Radiofrequency-Based Catheter Ablation for Treating Ventricular Arrhythmias Arising From the Papillary Muscles of the Left Ventricle, Guided by Intracardiac Echocardiography and Image Integration. Circ Arrhythm Electrophysiol. 2016 Apr;9(4):e003874. doi: 10.1161/CIRCEP.115.003874. PMID 27069089